CLINICAL TRIAL: NCT03513055
Title: Influence of Injection Technique of Premixed Insulin on Glucose Excursion in Type 2 Diabetes Mellitus Using CGMS
Brief Title: Influence of Injection Technique of Premixed Insulin on Glucose Excursion in Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENDO20180205-06
Record Dates: First submitted 2018-04-17; First posted 2018-05-01 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Type2 Diabetes Mellitus
Keywords: glucose excursions; insulin technique; insulin antibodies; premixed insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- inject premixed insulin (Experimental): patients inject premixed insulin themselves then nurse inject premixed insulin
  Interventions: Other: nurse inject premixed insulin

INTERVENTIONS:
Other: nurse inject premixed insulin — nurse inject premixed insulin，coaching in the injection technique

SUMMARY:
To compare patients and nurses using insulin pen injector to inject premixed insulin respectively, using continuous glucose monitoring system to evaluate the glucose excursion in the two sets, study the relationship between glucose excursion and inject technique in type 2 diabetes mellitus.

DETAILED DESCRIPTION:
A total of 60 patients with type 2 diabetes who used premixed insulin will enrolled in this study.Measure their blood pressure，height and weight, BMI, liver and kidney function, blood lipids, glycosylated hemoglobin, fasting glucose, 2 hour postprandial glucose，fasting C peptide, 2 hour postprandial C peptide, fasting glucagon, 2 hour postprandial glucagon,fasting serum insulin，2 hour postprandial serum insulin，urinary albumin and insulin antibodies.The first and second days，the patients inject premixed insulin themselves，the specialist nurse graded the patient's injection technique score.The third and the fourth days the nurse change a new insulin with the same types maintain the same injection dosage.The patient need perform continuous glucose monitoring system(CGMS) for 96-hours.

ELIGIBILITY:
Inclusion Criteria:

1. type 2 diabetes patients
2. aged 20-80 years
3. had been on premixed insulin and used an insulin pen for at least 3 months
4. fasting glucose between 6.1-16 mmolL, postprandial(or random) glucose below 22.2mmol/L.
5. No acute complications such as diabetic ketoacidosis, diabetic hypertosmolar syndrome.
6. Subjects were able and willing to ues CGMS and eat regularly.
7. Patients who were able to inject insulin themselves or actual injections can be accompanied.

Exclusion Criteria:

1. Insulin allergy.
2. There has been a history of drug abuse and alcohol dependence in the past five years, or systemic hormone therapy within 3 months.
3. Patients with poor compliance and irregular eating and exercise.
4. Infection or stress within four weeks.
5. Patients unable to tolerate CGMS.
6. patients with pregnancy, breast-feeding, planning to have a baby
7. patients with coagulopathy, serious complication,such as cardiovascular disease, end stage renal disease; and patients with severe retinopathy or other eye problems that impair their visual function, or cognitive dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-05-07 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint was the relationship between MAGE and injection score | 6 DAYS
  the relationship between the 24-h mean amplitude of glycemic excursions (MAGE) and injection score
the relationship between HbA1C and injection score | 6 DAYS
  the relationship between HbA1C and injection score
the relationship between SDBG and injection score | 6 DAYS
  the relationship between SDBG and injection score

SECONDARY OUTCOMES:
the relation between insulin antibodies and glucose excursions | 6 DAYS
  the 24-h mean amplitude of glycemic excursions (MAGE)

CONTACTS AND LOCATIONS:
Overall Officials: YUAN LU, master, Study Director — Nanjing Medical University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yuan L, Li F, Jing T, Ding B, Luo Y, Sun R, Wang X, Diao H, Su X, Ye L, Ma J. Insulin Injection Technique is Associated with Glycemic Variability in Patients with Type 2 Diabetes. Diabetes Ther. 2018 Dec;9(6):2347-2356. doi: 10.1007/s13300-018-0522-1. Epub 2018 Oct 19. PMID 30341664